CLINICAL TRIAL: NCT03763864
Title: Développement de Tests Fonctionnels in Vitro à Partir de Cellules Primaires de Patients Atteints de Maladies Monogéniques
Brief Title: Development of In Vitro Functional Assays From Primary Cells of Patients With Monogenic Diseases
Acronym: OPERANDO
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Apteeus (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APTEEUS001
Record Dates: First submitted 2018-11-29; First posted 2018-12-04 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Monogenic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inherited disorders (Other)
  Interventions: Other: Skin Biopsy

INTERVENTIONS:
Other: Skin Biopsy — Skin Biopsy

SUMMARY:
The objective of this project is to build a collection of biological samples consisting of fibroblasts and primary keratinocytes from patients with orphan monogenic diseases and to use these cells in the customization of functional tests. The miniaturized tests we are setting up make it possible to distinguish patient cells from control cells. They can be used to test molecules or for the development of diagnostic tests.

As part of the research protocol, the investigating physicians will be able to perform a skin biopsy on their patient included in the study. APTEEUS will isolate fibroblasts and keratinocytes and ensure their preservation. As part of the project, it is planned to preserve the biological samples collected and to preserve the collection after the end of the study. Skin fibroblasts and keratinocytes that are isolated from the biopsy are cells that can be preserved and amplified. They are a material of choice for the functional study of many monogenic diseases.

This study will allow the adaptation of tools dedicated to the functional study of monogenic diseases in order to help in the research and development of new treatments for these diseases, but also to highlight and explain the inter-individual variability of symptoms and responses to treatments, and finally, to help in the development of diagnostic methods.

Patients with orphan monogenic diseases whose genetic defect has been confirmed and for whom the study of the disease can be performed on fibroblasts, keratinocytes or cells derived from them, may be included in the study. Subjects, after information and consent, will undergo a skin biopsy. The sample will be sent directly to the promoter company APTEEUS, which will carry out all in vitro developments. The fibroblasts and keratinocytes will be preserved and will constitute a collection of cells "orphan monogenic diseases". The samples can be reused for new research in the same field.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an orphan monogenic disease (without any satisfactory therapeutic option).
* Patients with a pathology whose functional cause can be demonstrated by APTEEUS technologies in skin cells or cells derived from them.

Exclusion Criteria:

* Patients whose molecular cause is not clearly identified.
* Patients contraindicated for skin biopsy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-09-06 (Actual); Primary Completion 2025-09-06 (Estimated); Study Completion 2025-09-06 (Estimated)

PRIMARY OUTCOMES:
Measurement of the residual enzymatic activity on the isolated fibroblast and or keratinocytes using appropriate methodology. | 6 months
  The function of the impaired enzyme will be assessed by measuring in vitro the residual enzymatic activity using labeled substrate. Technologies used are based on mass spectrometry. Residual enzymatic activity will be expressed as a percentage of normal controls.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU, Lille, France